CLINICAL TRIAL: NCT03788252
Title: RolE of AST120 in sarCOpenia preVEntion in pRe-dialYsis Chronic Kidney Disease Patients (RECOVERY): Prospective Open-label Randomized Controlled Multicenter Study
Brief Title: Role of AST120 for Sarcopenia Prevention in Pre-dialysis Chronic Kidney Disease
Acronym: RECOVERY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gumi Cha Medical Center (Other)
Responsible Party: Principal Investigator, Jun Chul Kim, Professor, Gumi Cha Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GM18-11
Record Dates: First submitted 2018-11-28; First posted 2018-12-27 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Sarcopenia; AST-120; Indoxyl sulfate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Renamezin (AST-120) group or non-Renamezin group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renamezin (Active Comparator): oral treatment duration: three times a day, 7 capsules (2g) once, for 48 weeks
  Interventions: Drug: Renamezin
- Non-Renamezin (No Intervention): no use of Renamezin

INTERVENTIONS:
Drug: Renamezin — 7 capsules once, three times a day, for 48 weeks
  Other Names: Renamezin administration
  Arms: Renamezin

SUMMARY:
This study is to assess the effect of 48 weeks administration of Renamezin capsule on prevention of sarcopenia in pre-dialysis patients with chronic kidney disease.

DETAILED DESCRIPTION:
Skeletal muscle atrophy, referred to as sarcopenia, and impaired physical performance are accompanied in chronic kidney disease patients during disease progression. Decreased physical performance derived from sarcopenia precipitates poor prognostic influence in the clinical outcome, as reported in previous studies showing correlations between poor physical performance, poor quality of life, poor renal prognosis, and mortality. Therefore, maintaining physical performance is mandatory to improve the prognosis of chronic kidney disease patients.

AST-120 is an oral absorbent capsule designed to remove circulating indoxyl sulfate, a uremic toxin. As indoxyl sulfate is reported to cause mitochondrial dysfunction in skeletal muscle, AST-120 contributes to the recovery of mitochondrial function by reducing indoxyl sulfate. In addition, AST-120 is reported to delay the initiation of dialysis and the decrease of glomerular filtration rate and the increase of serum creatinine level. However, the effect of AST-120 on sarcopenia in pre-dialysis patients have not been reported. This study is to investigate the effect of AST-120 on sarcopenia prevention in pre-dialysis chronic kidney disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult older than 19 years
* Pre-dialysis chronic kidney disease
* Serum creatinine level 2.0-5.0 mg/dL or MDRD or CKD-EPI eGFR 15-60 mL/min/1.73 m²
* Serum albumin ≥ 3.0 g/dL
* No previous use of oral absorbant during 4 weeks prior to screening
* No change of treatment for chronic kidney disease during 4 weeks prior to screening
* Written informed consent to participate in this clinical study
* Capable of independent physical activity, an assisted device use is acceptable

Exclusion Criteria:

* Impaired GI peristalsis
* Uncontrolled constipation
* Prior renal transplant
* On immunosuppressant (small dose users may be accepted according to the PI's decision)
* GI ulcer or esophageal varix
* Uncontrolled hypertension (systolic BP ≥180 mmHg or diastolic BP ≥110 mmHg)
* History of admission for an acute cardiovascular incident within 3 months prior to screening
* Current acute infection state
* Liver function failure (ALT, AST over 2.5 times of normal reference range)
* Uncontrolled diabetes patient (HbA1c >10 % or fasting glucose >250 mg/dL)
* Malignancy (patients of post-remission 5 years without any recurrence can be enrolled, except for squamous cell carcinoma in situ)
* Pregnancy, on breastfeeding
* Not agreed to medical contraceptive use during participating in the study
* Concurrent participation in another clinical trial
* Drug or alcohol-dependent
* Other clinical trial medication administration more than once within 30 days prior to enrollment
* Expected dialysis or kidney transplantation within 3 months prior to enrollment
* Dependent physical activity
* Musculoskeletal disease that may debilitate functional independence
* Lower limb amputee not using a prosthesis
* Severe retinal disease (e.g., proliferative diabetic retinopathy, vitreous hemorrhage)
* Claudication
* Other patients inappropriate to participate by the PI's decision

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Change of 6 meter walking speed at 24 weeks | Change of baseline 6 meter walking speed at 24 weeks
  As a measure of physical performance, 6 meter walking test is used. Static start and dynamic start speed will be assessed twice each.
Change of 6 meter walking speed at 48 weeks | Change of baseline 6 meter walking speed at 48 weeks
  As a measure of physical performance, 6 meter walking test is used. Static start and dynamic start speed will be assessed twice each.

SECONDARY OUTCOMES:
Body composition test | Baseline, 24 week, 48 week
  Bioelectrical impedance analysis (using InBody S10)
Serum level of indoxyl sulfate, myostatin, Tumor Necrosis Factor-alpha, Interleukin-6 | Baseline, 24 week, 48 week
  Level of serum indoxyl sulfate, myostatin, TNF-alpha, and IL-6 will be obtained by laboratory blood test.
Serum level of creatinine and estimated Glomerular Filtration Rate (eGFR) | Baseline, 24 week, 48 week
  Level of serum creatinine, and eGFR (mL/min/1.73 m²) will be obtained by laboratory blood test.
Kidney Disease Quality of Life Short Form 1.3 (KDQOL-SF 1.3) | Baseline, 24 week, 48 week
  Health-related quality of life (HRQOL) is assessed via KDQOL-SF 1.3. KDQOL-SF 1.3 is validated questionnaires to assess HRQOL. HRQOL consists of three subscales; physical health, mental health, and kidney disease health. The summation of subscales ranges between 0 - 100, and the higher values indicate the better HRQOL status.
Charlson Co-morbidity Index | Baseline, 24 week, 48 week
  Charlson Co-morbidity Index is used to assess underlying co-morbidity of each patient. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use. Age weighting is added to total comorbidity score in a score of zero to four.
International Physical Activity Questionnaire Short Form | Baseline, 24 week, 48 week
  International Physical Activity Questionnaire (IPAQ) Short Form is used to assess the amount of time spent for daily physical activity. IPAQ Short Form comprises of 7 questionnaires of activities which asks to report time spent for each activity during last week.
Grip strength | Baseline, 24 week, 48 week
  Using TAKEI handgrip strength dynamometer (TKK5401, Japan), grip strength while flexing elbow and extending elbow will be assessed.
24h body activity measure | Baseline, 24 week, 48 week
  Using BAND2 model of InBody cooperation, activity amount of each participant is collected for 7 days.

OTHER OUTCOMES:
Time of dialysis initiation | Through study completion, an average of 2 years
  If a patient requires dialysis initiation during study period, the date is recorded.
Rate of hospital admission | Through study completion, an average of 2 years
  The rate of patients requiring in-patient care during the study participation is calculated.
Death rate | Through study completion, an average of 2 years
  Death rate is calculated if any patients expire during participation.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chul Kim, MD, PhD, Principal Investigator — CHA Gumi Medical Center
Locations (1):
- CHA Gumi Medical Center, Gumi, Gyeongsangbuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee SM, Han MY, Kim SH, Cha RH, Kang SH, Kim JC, An WS. Indoxyl Sulfate Might Play a Role in Sarcopenia, While Myostatin Is an Indicator of Muscle Mass in Patients with Chronic Kidney Disease: Analysis from the RECOVERY Study. Toxins (Basel). 2022 Sep 23;14(10):660. doi: 10.3390/toxins14100660. PMID 36287929
- [Derived] Shin J, Kim JC, Kim SH. Reply - Letter to the editor: Comment on "phase angle as a marker for muscle health and quality of life in patients with chronic kidney disease". Clin Nutr. 2022 Sep;41(9):2058. doi: 10.1016/j.clnu.2022.07.020. Epub 2022 Jul 21. No abstract available. PMID 35963741
- [Derived] Cha RH, Kang SH, Han MY, An WS, Kim SH, Kim JC. Effects of AST-120 on muscle health and quality of life in chronic kidney disease patients: results of RECOVERY study. J Cachexia Sarcopenia Muscle. 2022 Feb;13(1):397-408. doi: 10.1002/jcsm.12874. Epub 2021 Dec 3. PMID 34862753